CLINICAL TRIAL: NCT06627998
Title: Study of the Prevalence of Osteo-metabolic Complications in Patients With Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Giustina, Professor of Endocrinology, IRCCS San Raffaele
Other Study IDs: OsteoTIR
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Cancer of Thyroid; Vertebral Fracture; Osteoporosis
MeSH Terms: conditions — Thyroid Neoplasms; Spinal Fractures; Osteoporosis | interventions — Diagnosis; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic (chest x-ray /DXA)and clinical data collected for clinical practice — Biochemical, clinical and radiological data performed for clinical practice will be retrospectively collected. Osteoporosis and vertebral fractures will be diagnosed through DXA scan and vertebral morphometry.

SUMMARY:
This is a multicenter retrospective observational study aimed to evaluate the prevalence of osteo-metabolic complications in patients with thyroid cancer.

DETAILED DESCRIPTION:
Approximately 150-200 outpatients evaluated in the Endocrinology Unit of the IRCCS San Raffaele Hospital and the Nuclear Medicine Unit of the Spedali Civili of Brescia will be included in the study.

During the follow-up visits, patients who meet the inclusion criteria will be offered inclusion in the study. After signing the informed consent, the patient's anamnestic and clinical (biochemical, radiological, anamnestic) data will be retrospectively collected in an electronic database. Sensitive data will be anonymized.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Histological diagnosis of Thyroid Carcinoma
* radiological data from chest x-ray in lateral projection in the preoperative evaluation on which the vertebral morphometry
* Signing of the informed consent

Exclusion Criteria:

* Subjects not falling within the previously described criteria are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid cancers who have been evaluated at the outpatient clinics of the Endocrinology Unit of the IRCCS San Raffaele Hospital and the Nuclear Medicine Unit of the Spedali Civili di Brescia.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the incidence and prevalence of osteoporosis and vertebral fractures in Patients With Thyroid Cancer | 1 year
  To estimate the incidence and prevalence of osteoporosis and vertebral fractures detected through DXA scan and vertebral morphometry. The effects on bone complications of the patients' clinical and biochemical characteristics will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Giustina, Milan, Italy